CLINICAL TRIAL: NCT02464293
Title: A Pilot Evaluation of Mindfulness-based Cognitive Therapy for People With Huntington's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster University (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Dr Jane Simpson, Research Director, Doctorate in Clinical Psychology, Lancaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHDN Seed Fund Project 561; 15/NW/0238 (Other: NHS National Research Ethics Service REC)
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Huntington Disease
Keywords: depression; anxiety; stress
MeSH Terms: conditions — Huntington Disease; Depression; Anxiety Disorders | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mindfulness-based cognitive therapy (Experimental)
  Interventions: Other: Mindfulness-based cognitive therapy

INTERVENTIONS:
Other: Mindfulness-based cognitive therapy — An 8 week course of mindfulness-based cognitive therapy

SUMMARY:
This is a pilot study to see whether mindfulness-based cognitive therapy, which is a type of psychological therapy, is able to improve the psychological wellbeing of people who have the gene for Huntington's disease.

DETAILED DESCRIPTION:
Huntingdon's disease (HD) is a genetic neurodegenerative condition which causes problems with movement, coordination and cognitive functioning, and emotional difficulties are also commonly experienced. It is believed to affect around five to ten in 100,000 people of European descent, with recent UK estimates as high as 11.2-13.5. Each child of an affected person has a 50% chance of inheriting the condition. As age of diagnosis is typically around 35-55, with time from diagnosis to death around 20 years, those who are diagnosed have often seen their parents affected by the condition.

Many people at various stages of HD (including those who carry the gene but are pre-symptomatic) experience low mood, anxiety and other psychological difficulties. Indeed, alongside functional capacity, mood may be one of the main factors which contributes to health related quality of life, more so than discrete motor problems, or cognitive impairment. In addition, reports from patients suggest emotional and social concerns are important for individuals with the condition at the pre-symptomatic stage, and these concerns remain throughout the disease course. Medication may be effective to alleviate psychological difficulties for some people, but its efficacy has not been conclusively proven and it is not suitable for all. Psychological interventions may provide an alternative or additional way of alleviating distress.

Although it is commonly presumed that biological factors are the main determinants of psychological distress in people with HD, several studies have indicated that, while these may indeed be important, psychological factors are also significant. For example beliefs about the disease and coping mechanisms are associated with poorer mental health and higher levels of depression. Such psychological beliefs and coping patterns can be adaptively changed using psychological interventions, for example cognitive-based psychological therapies.

Little progress has been reported on the development of psychological interventions in HD despite the fact that people with HD have expressed an interest in psychological approaches and these are currently being successfully developed for people with other neurological conditions (e.g., in people with Parkinson's disease). It is therefore proposed to pilot mindfulness-based cognitive therapy (MBCT) which, although originally developed to help people with remitted depression from relapse, has been increasingly used to help people with current difficulties. It has also been piloted with people with Parkinson's disease who found it an acceptable intervention and reported improvements in self-management and psychological wellbeing. In general, MBCT has also recorded other gains including improved sleep quality and social functioning. It has also received sufficient evidence for it to be a recommended approach in the UK NICE guidelines for people with a history of depression. MBCT can also reduce anxiety and provides group support. There are also indications that mindfulness training can improve neurocognitive functioning, even in people with neurodegenerative disease. Finally, a psychological therapy subgroup within the European Huntington's Disease Network has recently been formed, thus indicating the rise of interest in psychological approaches and the timely nature of this work.

Hence this study will provide the first indication of whether MBCT, a therapeutic approach with an established evidence base, would be acceptable and useful for people with HD. In order to meet this aim, MBCT will be delivered to two groups, one to individuals who carry the gene but are pre-symptomatic and one to individuals who have begun to experience symptoms but are at an early stage of the disease course.

Approaches to outcome evaluation should be incremental, with lower cost studies, e.g., qualitative investigations and case studies, being conducted before investment in randomised controlled trials is considered. Thus this study will follow this guidance by collecting both qualitative and quantitative data. The qualitative data will be analysed using interpretative phenomenological analysis, a methodology previously used in other qualitative studies on MBCT. Semi-structured interviews will provide data on the acceptability of the intervention and detailed accounts of participants' experience after the intervention has been provided. This will inform whether the MBCT intervention needs to be changed or adapted in further trials. The quantitative data will be used to provide basic pre and post intervention comparisons on a number of outcome variables relevant to MBCT, with the hypothesis that performance on these measures will improve post training. These data will also be used to estimate effect sizes for further trials so that these are suitably powered.

Given the considerable physical, cognitive and emotional consequences of the disease, HD not only affects the person with HD, but also those with whom they live, even in the pre-clinical phase. Family members often become caregivers and can have a reduced quality of life as a result, including experiencing low mood themselves. In fact, caregiver burden and caregiver depression is associated with depression of the person with HD and, alongside motor disturbances, depression of the person with HD is one of the main predictors of caregiver burden. Partners of people with HD can also experience reduced satisfaction with their relationship, sometimes more so than the person with HD themselves.

Thus this study will also investigate the views of a family member (e.g. partner, parent, child) of the person participating in the intervention. As the intervention is aimed at alleviating psychological distress in the person with HD, it is hypothesised that this in turn will also have an effect on the family member's wellbeing. Also, higher levels of mindfulness are associated with higher levels of satisfaction in partner relationships, perhaps due to more adaptive conflict resolution and better emotional recognition and management. Participants in MBCT have reported increased empathy and perspective taking, being more able to respond mindfully in relationships. Thus increased mindfulness of the person with HD may benefit family and social relationships.

In addition, caregivers' views about the symptoms or quality of life of the person with HD may not always match the person with HD themselves. Furthermore, certain symptom changes which are beneficial to the person with HD may not be so to the caregiver, and thus the caregiver can offer an alternative perspective of the wellbeing (including behavioural and psychological changes) of the person with HD.

Both qualitative and quantitative data will be collected from a family member or close friend of the person with HD, where such a person is available and willing to take part. Semi-structured interviews with the family member will explore their perceptions on the acceptability of the intervention and experiences of the person with HD, as well as the impact on the family member personally and the wider family system. Data collected pre and post the intervention will assess any changes in their psychological wellbeing, caregiver burden and family relationships, with the hypothesis that wellbeing and relationships will improve post training and caregiver burden will decrease.

ELIGIBILITY:
Inclusion Criteria:

For those with HD:

Patient at Manchester Centre for Genomic Medicine (UK)

* All participants will have had genetic testing and shown to have the requisite CAG expansion on the huntingtin gene.
* Participants must be pre-symptomatic or at stage 1 (still able to function at home and at work and handle financial affairs)
* Clinical sign of depression (score on HADS of 7 or above)
* No significant medication changes in 6 weeks prior to starting the course

For those who are relatives or friends of those with HD:

* Must be a relative or friend of someone participating in the MBCT course

Exclusion Criteria:

* Active suicidal intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
depression post intervention | immediately post-intervention (up to two weeks afterwards)
  Change in Hospital Anxiety and Depression Scale (HADS) depression score pre to post intervention (People with HD only)
depression at 3 months | 3 months post-intervention
  Change in HADS depression score pre to 3 months post intervention
depression at 1 year | 1 year post-intervention
  Change in HADS depression score pre to 1 year post intervention

SECONDARY OUTCOMES:
depression mid-course | 4 weeks after start of intervention
  Change in HADS depression score pre to mid-course (4 weeks after start) (people with HD only)
anxiety mid-course | 4 weeks after start of intervention
  Change in HADS anxiety score pre to mid-course (4 weeks after start) (people with HD only)
anxiety post intervention | immediately post-intervention (up to two weeks afterwards)
  Change in HADS anxiety score pre to post-intervention (people with HD only)
anxiety at 3 months | 3 months post-intervention
  Change in HADS anxiety score pre to 3 months post intervention
anxiety at 1 year | 1 year post-intervention
  Change in HADS anxiety score pre to 1 year post intervention
stress mid course | 4 weeks after start of intervention
  Change in Depression Anxiety and Stress Scale (DASS) stress score pre to mid-course (4 weeks after start) (people with HD only)
stress post intervention | immediately post-intervention (up to two weeks afterwards)
  Change in DASS stress score pre to post course (people with HD only)
stress at 3 months | 3 months post-intervention
  Change in DASS stress score pre to 3 months post intervention
stress at 1 year | 1 year post-intervention
  Change in DASS stress score pre to 1 year post intervention
mindfulness mid-course | 4 weeks after start of intervention
  Change in Five Factor Mindfulness Questionnaire (FFMQ) score pre to mid-course (4 weeks after start) (people with HD only)
mindfulness post intervention | immediately post-intervention (up to two weeks afterwards)
  Change in FFMQ score pre to post course (people with HD only)
mindfulness at 3 months | 3 months post-intervention
  Change in FFMQ score pre to 3 months post intervention
mindfulness at 1 year | 1 year post-intervention
  Change in FFMQ score pre to 1 year post intervention
sleep post intervention | immediately post-intervention (up to two weeks afterwards)
  Change in Pittsburgh Sleep Quality Index (PSQI) score pre to post course (people with HD only)
sleep at 3 months | 3 months post-intervention
  Change in PSQI score pre to 3 months post intervention (people with HD only)
sleep at 1 year | 1 year post-intervention
  Change in PSQI score pre to 1 year post intervention (people with HD only)
quality of life post intervention | immediately post-intervention (up to two weeks afterwards)
  Change in World Health Organisation Quality of Life BREF) score (WHOQOL) pre to post course (people with HD only)
quality of life at 3 months | 3 months post-intervention
  Change in WHOQOL score pre to 3 months post intervention
quality of life at 1 year | 1 year post-intervention
  Change in WHOQOL score pre to 1 year post intervention
positive affect post intervention | immediately post-intervention (up to two weeks afterwards)
  Change in Positive And Negative Affect Scale (PANAS) positive items score pre to post course (people with HD only)
positive affect at 3 months | 3 months post-intervention
  Change in PANAS positive items score pre to 3 months post intervention
positive affect at 1 year | 1 year post-intervention
  Change in PANAS positive items score pre to 1 year post intervention
coping post intervention | immediately post-intervention (up to two weeks afterwards)
  Change in brief COPE score pre to post course (people with HD only)
coping at 3 months | 3 months post-intervention
  Change in brief COPE score pre to 3 months post intervention
coping at 1 year | 1 year post-intervention
  Change in brief COPE score pre to 1 year post intervention
relationship satisfaction at 3 months | 3 months post-intervention
  Change in Relationship Assessment Scale (RAS) score pre to 3 months post intervention (relatives/friends only)
relationship satisfaction at 1 year | 1 year post-intervention
  Change in RAS score pre to 1 year post intervention (relatives/friends only)
carer burden at 3 months | 3 months post-intervention
  Change in carer burden inventory score pre to 3 months post intervention (relatives/friends only)
carer burden at 1 year | 1 year post-intervention
  Change in carer burden inventory score pre to 1 year post intervention (relatives/friends only)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Simpson, PhD, Principal Investigator — Lancaster University
Locations (1):
- Central Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Background] Arran N, Craufurd D, Simpson J. Illness perceptions, coping styles and psychological distress in adults with Huntington's disease. Psychol Health Med. 2014;19(2):169-79. doi: 10.1080/13548506.2013.802355. Epub 2013 Jun 14. PMID 23767964
- [Background] Kristjanson LJ, Aoun SM, Oldham L. Palliative care and support for people with neurodegenerative conditions and their carers. Int J Palliat Nurs. 2006 Aug;12(8):368-77. doi: 10.12968/ijpn.2006.12.8.368. PMID 17077795
- [Background] Aubeeluck A, Buchanan H. The Huntington's disease quality of life battery for carers: reliability and validity. Clin Genet. 2007 May;71(5):434-45. doi: 10.1111/j.1399-0004.2007.00784.x. PMID 17489849
- [Background] Aubeeluck AV, Buchanan H, Stupple EJ. 'All the burden on all the carers': exploring quality of life with family caregivers of Huntington's disease patients. Qual Life Res. 2012 Oct;21(8):1425-35. doi: 10.1007/s11136-011-0062-x. Epub 2011 Nov 13. PMID 22081218
- [Background] Banaszkiewicz K, Sitek EJ, Rudzinska M, Soltan W, Slawek J, Szczudlik A. Huntington's disease from the patient, caregiver and physician's perspectives: three sides of the same coin? J Neural Transm (Vienna). 2012 Nov;119(11):1361-5. doi: 10.1007/s00702-012-0787-x. Epub 2012 Mar 8. PMID 22398875
- [Background] Barnes S, Brown KW, Krusemark E, Campbell WK, Rogge RD. The role of mindfulness in romantic relationship satisfaction and responses to relationship stress. J Marital Fam Ther. 2007 Oct;33(4):482-500. doi: 10.1111/j.1752-0606.2007.00033.x. PMID 17935531
- [Background] Barnhofer T, Crane C, Hargus E, Amarasinghe M, Winder R, Williams JM. Mindfulness-based cognitive therapy as a treatment for chronic depression: A preliminary study. Behav Res Ther. 2009 May;47(5):366-73. doi: 10.1016/j.brat.2009.01.019. Epub 2009 Feb 5. PMID 19249017
- [Background] Bihari, J, Mullan, E. Relating Mindfully: A Qualitative Exploration of Changes in Relationships Through Mindfulness-Based Cognitive Therapy. Mindfulness 5(1): 46-59, 2014.
- [Background] Cairns V, Murray C. How do the features of mindfulness-based cognitive therapy contribute to positive therapeutic change? A meta-synthesis of qualitative studies. Behav Cogn Psychother. 2015 May;43(3):342-59. doi: 10.1017/S1352465813000945. Epub 2013 Nov 11. PMID 24229765
- [Background] Craufurd, D, Snowden, JS. Neuropsychiatry and Neuropsychology. In G Bates, SJ Tabrizi, L Jones (Eds.), Huntington's disease (4th ed., pp. 36-65). Oxford: Oxford University Press. (2014)
- [Background] Craufurd D, Thompson JC, Snowden JS. Behavioral changes in Huntington Disease. Neuropsychiatry Neuropsychol Behav Neurol. 2001 Oct-Dec;14(4):219-26. PMID 11725215
- [Background] Dobkin RD, Menza M, Allen LA, Gara MA, Mark MH, Tiu J, Bienfait KL, Friedman J. Cognitive-behavioral therapy for depression in Parkinson's disease: a randomized, controlled trial. Am J Psychiatry. 2011 Oct;168(10):1066-74. doi: 10.1176/appi.ajp.2011.10111669. Epub 2011 Jun 15. PMID 21676990
- [Background] Eisendrath SJ, Delucchi K, Bitner R, Fenimore P, Smit M, McLane M. Mindfulness-based cognitive therapy for treatment-resistant depression: a pilot study. Psychother Psychosom. 2008;77(5):319-20. doi: 10.1159/000142525. Epub 2008 Jul 4. No abstract available. PMID 18600038
- [Background] Evans SJ, Douglas I, Rawlins MD, Wexler NS, Tabrizi SJ, Smeeth L. Prevalence of adult Huntington's disease in the UK based on diagnoses recorded in general practice records. J Neurol Neurosurg Psychiatry. 2013 Oct;84(10):1156-60. doi: 10.1136/jnnp-2012-304636. Epub 2013 Mar 12. PMID 23482661
- [Background] Fitzpatrick L, Simpson J, Smith A. A qualitative analysis of mindfulness-based cognitive therapy (MBCT) in Parkinson's disease. Psychol Psychother. 2010 Jun;83(Pt 2):179-92. doi: 10.1348/147608309X471514. Epub 2009 Oct 19. PMID 19843353
- [Background] Griffiths K, Camic PM, Hutton JM. Participant experiences of a mindfulness-based cognitive therapy group for cardiac rehabilitation. J Health Psychol. 2009 Jul;14(5):675-81. doi: 10.1177/1359105309104911. PMID 19515682
- [Background] Helder DI, Kaptein AA, Van Kempen GM, Weinman J, Van Houwelingen HC, Roos RA. Living with Huntington's disease: Illness perceptions, coping mechanisms, and patients' well-being. Br J Health Psychol. 2002 Nov;7(Part 4):449-462. doi: 10.1348/135910702320645417. PMID 12614496
- [Background] Ho AK, Gilbert AS, Mason SL, Goodman AO, Barker RA. Health-related quality of life in Huntington's disease: Which factors matter most? Mov Disord. 2009 Mar 15;24(4):574-8. doi: 10.1002/mds.22412. PMID 19097181
- [Background] Ho AK, Hocaoglu MB; European Huntington's Disease Network Quality of Life Working Group. Impact of Huntington's across the entire disease spectrum: the phases and stages of disease from the patient perspective. Clin Genet. 2011 Sep;80(3):235-9. doi: 10.1111/j.1399-0004.2011.01748.x. Epub 2011 Aug 4. PMID 21736564
- [Background] Jha AP, Stanley EA, Kiyonaga A, Wong L, Gelfand L. Examining the protective effects of mindfulness training on working memory capacity and affective experience. Emotion. 2010 Feb;10(1):54-64. doi: 10.1037/a0018438. PMID 20141302
- [Background] Julien CL, Thompson JC, Wild S, Yardumian P, Snowden JS, Turner G, Craufurd D. Psychiatric disorders in preclinical Huntington's disease. J Neurol Neurosurg Psychiatry. 2007 Sep;78(9):939-43. doi: 10.1136/jnnp.2006.103309. Epub 2006 Dec 18. PMID 17178819
- [Background] Kaptein, A.A, Helder, DI, Scharloo, M, Van Kempen, GMJ, Weinman, J, Van Houwelingen, HJC, Roos, RAC. Illness perceptions and coping explain well-being in patients with Huntington's disease. Psychology & Health, 21(4): 431-446. (2006)
- [Background] Kaptein AA, Scharloo M, Helder DI, Snoei L, van Kempen GM, Weinman J, van Houwelingen JC, Roos RA. Quality of life in couples living with Huntington's disease: the role of patients' and partners' illness perceptions. Qual Life Res. 2007 Jun;16(5):793-801. doi: 10.1007/s11136-007-9194-4. Epub 2007 Mar 21. PMID 17375373
- [Background] Kay, C, Fisher, E, Hayden, MR. Epidemiology. In G. Bates, S. J. Tabrizi & L. Jones (Eds.), Huntington's disease (4th ed., pp. 131-164). Oxford: Oxford University Press. 2014.
- [Background] Lowit A, van Teijlingen ER. Avoidance as a strategy of (not) coping: qualitative interviews with carers of Huntington's Disease patients. BMC Fam Pract. 2005 Sep 14;6:38. doi: 10.1186/1471-2296-6-38. PMID 16162290
- [Background] Ma SH, Teasdale JD. Mindfulness-based cognitive therapy for depression: replication and exploration of differential relapse prevention effects. J Consult Clin Psychol. 2004 Feb;72(1):31-40. doi: 10.1037/0022-006X.72.1.31. PMID 14756612
- [Background] Marciniak R, Sheardova K, Cermakova P, Hudecek D, Sumec R, Hort J. Effect of meditation on cognitive functions in context of aging and neurodegenerative diseases. Front Behav Neurosci. 2014 Jan 27;8:17. doi: 10.3389/fnbeh.2014.00017. eCollection 2014. PMID 24478663
- [Background] McCabe MP, Firth L, O'Connor E. A comparison of mood and quality of life among people with progressive neurological illnesses and their caregivers. J Clin Psychol Med Settings. 2009 Dec;16(4):355-62. doi: 10.1007/s10880-009-9168-5. Epub 2009 Jul 29. PMID 19639395
- [Background] Mestre TA, Ferreira JJ. An evidence-based approach in the treatment of Huntington's disease. Parkinsonism Relat Disord. 2012 May;18(4):316-20. doi: 10.1016/j.parkreldis.2011.10.021. Epub 2011 Dec 16. PMID 22177624
- [Background] Newberg AB, Serruya M, Wintering N, Moss AS, Reibel D, Monti DA. Meditation and neurodegenerative diseases. Ann N Y Acad Sci. 2014 Jan;1307:112-123. doi: 10.1111/nyas.12187. Epub 2013 Aug 7. PMID 23924172
- [Background] O'Connor EJ, McCabe MP. Predictors of quality of life in carers for people with a progressive neurological illness: a longitudinal study. Qual Life Res. 2011 Jun;20(5):703-11. doi: 10.1007/s11136-010-9804-4. Epub 2010 Dec 2. PMID 21127997
- [Background] Paulsen JS, Ready RE, Hamilton JM, Mega MS, Cummings JL. Neuropsychiatric aspects of Huntington's disease. J Neurol Neurosurg Psychiatry. 2001 Sep;71(3):310-4. doi: 10.1136/jnnp.71.3.310. PMID 11511702
- [Background] Pickett T, Altmaier E, Paulsen, JS. Caregiver burden in Huntington's disease. Rehabilitation Psychology 52(3): 311-318. 2007.
- [Background] Read J, Jones R, Owen G, Leavitt BR, Coleman A, Roos RA, Dumas EM, Durr A, Justo D, Say M, Stout JC, Tabrizi SJ, Craufurd D; TRACK-HD investigators. Quality of life in Huntington's disease: a comparative study investigating the impact for those with pre-manifest and early manifest disease, and their partners. J Huntingtons Dis. 2013;2(2):159-75. doi: 10.3233/JHD-130051. PMID 25063513
- [Background] Ready RE, Mathews M, Leserman A, Paulsen JS. Patient and caregiver quality of life in Huntington's disease. Mov Disord. 2008 Apr 15;23(5):721-6. doi: 10.1002/mds.21920. PMID 18175350
- [Background] Ree MJ, Craigie M A. Outcomes following mindfulness-based cognitive therapy in a heterogeneous sample of adult outpatients. Behavior Change 24(2): 70-86, 2007.
- [Background] Smith JA. Interpretative phenomenological analysis : theory, method and research. London: Sage. 2009.
- [Background] Spinney L. Uncovering the true prevalence of Huntington's disease. Lancet Neurol. 2010 Aug;9(8):760-1. doi: 10.1016/S1474-4422(10)70160-5. Epub 2010 Jun 30. No abstract available. PMID 20594915
- [Background] Splevins K, Smith A, Simpson J. Do improvements in emotional distress correlate with becoming more mindful? A study of older adults. Aging Ment Health. 2009 May;13(3):328-35. doi: 10.1080/13607860802459807. PMID 19484596
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] Teasdale JD, Williams JMG, Segal, ZV. The Mindful Way Workbook: An 8-week Program to Free Yourself from Depression and Emotional Distress. New York, New York: Guildford Press. 2014.
- [Background] Videnovic A. Treatment of huntington disease. Curr Treat Options Neurol. 2013 Aug;15(4):424-38. doi: 10.1007/s11940-013-0219-8. PMID 23417276
- [Background] Wachs K, Cordova JV. Mindful relating: exploring mindfulness and emotion repertoires in intimate relationships. J Marital Fam Ther. 2007 Oct;33(4):464-81. doi: 10.1111/j.1752-0606.2007.00032.x. PMID 17935530
- [Background] Williams JK, Hamilton R, Nehl C, McGonigal-Kenney M, Schutte DL, Sparbel K, Birrer E, Tripp-Reimer T, Friedrich R, Penziner E, Jarmon L, Paulsen J. "No one else sees the difference: "family members' perceptions of changes in persons with preclinical Huntington disease. Am J Med Genet B Neuropsychiatr Genet. 2007 Jul 5;144B(5):636-41. doi: 10.1002/ajmg.b.30479. PMID 17219384
- [Background] Williams JK, Skirton H, Paulsen JS, Tripp-Reimer T, Jarmon L, McGonigal Kenney M, Birrer E, Hennig BL, Honeyford J. The emotional experiences of family carers in Huntington disease. J Adv Nurs. 2009 Apr;65(4):789-98. doi: 10.1111/j.1365-2648.2008.04946.x. Epub 2009 Feb 9. PMID 19228233
- [Background] Winbush NY, Gross CR, Kreitzer MJ. The effects of mindfulness-based stress reduction on sleep disturbance: a systematic review. Explore (NY). 2007 Nov-Dec;3(6):585-91. doi: 10.1016/j.explore.2007.08.003. PMID 18005910
- [Derived] Eccles FJR, Craufurd D, Smith A, Davies R, Glenny K, Homberger M, Peeren S, Rogers D, Rose L, Skitt Z, Theed R, Simpson J. A feasibility investigation of mindfulness-based cognitive therapy for people with Huntington's disease. Pilot Feasibility Stud. 2020 Jun 24;6:90. doi: 10.1186/s40814-020-00631-z. eCollection 2020. PMID 32595978
- See also: Medical Research Council. (2008). Developing and evaluating complex interventions: new guidance. — http://www.mrc.ac.uk/Utilities/Documentrecord/index.htm?d=MRC004871